CLINICAL TRIAL: NCT00143039
Title: Amniotic Fluid Tandem Mass Spectrometry for Pregnancies Complicated by Nonimmune Hydrops and Severe Symmetrical Intrauterine Growth Restriction-A Multicenter Prospective Pilot Cohort Study
Brief Title: Amniotic Fluid Tandem Mass Spectrometry for Pregnancies Complicated by NIH and Severe Symmetrical IUGR
Acronym: TandemMS
Status: Terminated | Type: Observational
Why Stopped: No metabolic disordered ID'd by TMS in either control/test group at >50%enrolled
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Other Study IDs: OBX 0005.3; Tandem MS - 0005.3
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Hydrops Fetalis; Fetal Growth Retardation
Keywords: NIH; Severe Symmetrical IUGR; Tandem Mass Spectrometry; Nonimmune Hydrops; Severe Symmetrical Intrauterine Growth Restriction
MeSH Terms: conditions — Hydrops Fetalis; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NIH/SSIUGR fetuses: Group 1 includes pregnancies complicated by a fetus with either Non-Immune Hydrops or Severe Symmetrical IUGR.
  Interventions: Procedure: Tandem MS test for inborn errors of metabolism
- Control-Normal fetus: Group 2 includes all normally appearing fetuses on U/S who will be having a diagnostic amniocentesis as part of their routine care.
  Interventions: Procedure: Tandem MS test for inborn errors of metabolism

INTERVENTIONS:
Procedure: Tandem MS test for inborn errors of metabolism — Tandem MS spectrometry test will be done on all maternal blood, amniotic fluid and newborn blood samples for both groups.
  Other Names: Tandem MS

SUMMARY:
The objective of this pilot study is to prospectively evaluate amniotic fluid of pregnancies complicated by non-immune hydrops and severe symmetrical intrauterine growth restriction by tandem mass spectrometry for inborn errors of metabolism.

DETAILED DESCRIPTION:
Nonimmune hydrops (NIH) and severe symmetrical intrauterine growth restriction (IUGR) represent two obstetrical circumstances that occur with relative frequency yet often escape adequate etiology assessment and diagnosis prior to and after birth. Both of these conditions have high perinatal and neonatal mortality rates. While antepartum ultrasound and amniotic fluid evaluations of fetal karyotype and viral DNA studies diagnose some etiologies for NIH and severe symmetrical IUGR, large percentages of NIH (30-40%) and IUGR (20-30%) cases are attributed to idiopathic causes. Because of this uncertainty in diagnosis, many cases are subjected to prolonged antepartum hospitalization with intensive fetal monitoring and urgent delivery by Cesarean section for non-reassuring fetal status, only to succumb to a neonatal demise in the nursery. A small percentage (1-2%) of these cases are found to be due to inborn errors of metabolism by neonatal and/or postmortem evaluation; however, when combined together, greater than 50% of NIH and IUGR cases have no identifiable etiology. Therefore, any new test that may make a diagnosis for NIH or severe symmetrical IUGR prior to delivery would be extremely important to the management of both the mother and the infant. Tandem mass spectrometry for inborn errors of metabolism may represent a new tool for assessing, identifying, and treating currently unexplained cases of NIH and severe symmetrical IUGR.

This is a prospective pilot cohort study of all pregnancies complicated by NIH and severe symmetrical IUGR within the Pediatrix-Obstetrix network. This network encompasses several perinatal sites throughout the United States with corresponding neonatal intensive care units utilizing a computerized patient database (RDS). The objective of this study is to prospectively evaluate amniotic fluid of pregnancies complicated by NIH and severe symmetrical IUGR by a method called tandem mass spectrometry for inborn errors of metabolism.

ELIGIBILITY:
NIH Inclusion Criteria:

* Singleton gestation
* 18 years of age or older
* Excess extracellular fluid in at least two fetal sites as noted by ultrasound: abdomen (ascites), the chest (pleural and pericardial effusions), the skin (edema > 5mm), the amniotic cavity (polyhydramnios), and the placenta (thickening > 6cm)
* NIH diagnosis > 15w0d gestation
* Diagnostic amniocentesis performed at > 15w0d gestation

NIH Exclusion Criteria:

* Immune-mediated hydrops fetalis as diagnosed by maternal red cell antigens and fetal anemia suspected by middle cerebral artery doppler ultrasound and/or confirmed by percutaneous umbilical blood sampling
* Structural anomaly identified by ultrasound
* Chromosomal aneuploidy
* Multiple gestations

IUGR Inclusion Criteria:

* Singleton gestation
* 18 years of age or older
* Severe symmetrical IUGR defined as a > 3 week lag of all fetal ultrasound measurements (biparietal diameter, head circumference, abdominal circumference, and femur length)
* IUGR diagnosis between 24-32 weeks gestation
* Diagnostic amniocentesis performed prior to 32 weeks gestation

IUGR Exclusion Criteria:

* Asymmetrical IUGR
* Structural anomaly identified by ultrasound
* Chromosomal aneuploidy
* Multiple gestations

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnancies complicated by NIH or SSIUGR fetuses as compared to a control group of pregnancies with normally appearing fetuses requiring a diagnostic amniocentesis as part of her care.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2006-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Will assess whether amniotic fluid tandem mass spectrometry results are valid when compared to neonatal blood samples for normal pregnancies and those pregnancies complicated by NIH and severe symmetrical IUGR. | comparrison down with in 2 days of life.
  Will assess whether amniotic fluid tandem mass spectrometry results are valid when compared to neonatal blood samples for normal pregnancies and those pregnancies complicated by NIH and severe symmetrical IUGR.

SECONDARY OUTCOMES:
Incidence of Neonatal Complications | during the neonatal period
  Will include neonatal complications in pregnancies complicated by NIH and severe symmetrical IUGR.

CONTACTS AND LOCATIONS:
Overall Officials: Karrie Francois, MD, Principal Investigator — Pediatrix-Obstetrix Medical Group, Inc.
Locations (11):
- United States (11):
  - Banner Good Sammaritan Hospital, Phoenix, Arizona
  - Banner Desert Samaritan Hospital, Phoenix, Arizona
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Good Samaritan Hospital, San Jose, California
  - Swedish Medical Center, Denver, Colorado
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - DeKalb Medical Center, Decatur, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - Swedish Medical Center, Seattle, Washington